CLINICAL TRIAL: NCT02105597
Title: A Smartphone Application to Improve Medication Adherence Among People With Type 2 Diabetes Mellitus in Singapore: A Randomized Controlled Trial
Brief Title: A Smartphone Application to Improve Medication Adherence Among People With Type 2 Diabetes Mellitus in Singapore
Acronym: iADHERE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor patient recruitment
Sponsor: Singapore General Hospital (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: iADHERE-01
Record Dates: First submitted 2014-03-28; First posted 2014-04-07 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; Medication adherence; Compliance; Mobile health
MeSH Terms: conditions — Diabetes Mellitus; Medication Adherence; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile application (Experimental)
  Interventions: Other: Mobile application
- Standard care (No Intervention)

INTERVENTIONS:
Other: Mobile application — The intervention in this study is a mobile application which will be downloaded into the participant's smartphone.
  Arms: Mobile application

SUMMARY:
Background: Diabetes mellitus (DM) is a major cause of morbidity and mortality worldwide. Long-term glycemic control is important to prevent or delay the onset of DM related complications. Patients often fail to achieve optimal glycemic control from pharmacotherapy due to non-adherence. With the high prevalence of smartphone usage locally and among the developed countries, there has been a growing interest to deliver interventions through mobile applications. In this study, a mobile application targeted at improving medication adherence among people with Type 2 DM will be developed and evaluated.

Aims: This study aims to (i) design a smartphone application to improve medication adherence and (ii) evaluate its impact on clinical outcomes, health-related quality of life (HRQoL) and health status among patients with Type 2 DM.

Hypothesis: The use of a smartphone application can improve medication adherence among patients with Type 2 DM, as well as clinical outcomes, HRQoL and health status.

Methods: This is a randomized, open-label controlled trial involving patients with Type 2 DM managed at Singapore General Hospital. Patients seen at the institution's Diabetes Centre and those referred to the pharmacist-led Medication Therapy Management service are eligible to participate. Patients in the intervention group will have the mobile application downloaded onto their smartphones, while those in the control group will receive the usual standard of care. The primary outcome will be change in self-reported medication adherence, determined using the 8-item Morisky Medication Adherence Scale. Secondary outcomes include change in HbA1c, blood glucose, frequency of dose titrations, addition or removal of oral hypoglycemic agents, HRQoL (measured using the Audit of Diabetes Dependent Quality of Life) and health status (measured using the EuroQol-5D-5L and EuroQol Visual Analogue Scale). All outcomes will be measured at baseline and at the end of the 6-month study period (± 4 weeks).

Significance: The development and evaluation of a mobile application to improve adherence among patients with Type 2 DM in Singapore is the first of its kind, and the findings of this study will provide the much-needed evidence to demonstrate the effectiveness of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Existing Type 2 DM managed at SGH Diabetes Centre and those referred to the pharmacist-led MTM service
* Age≥ 40 years
* HbA1c≥ 8.0
* Suspected non-adherence (e.g. admitted to have missed doses, HbA1c not at target despite frequent dose titrations, recent DM related hospitalization/ emergency visit)
* Owns a iOS smartphone with Wi-Fi or data plan

Exclusion Criteria:

* Unable to manage own medications (e.g. taken care of by caregiver, nursing home patients, cognitive impairment)
* Unable to read and comprehend English
* Physical impairment that precludes the use of smart phone functions (e.g. deformed finger joints, amputation)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported medication adherence | Baseline (at recruitment) and 6 months (+/- 4 weeks)
  Self-reported medication adherence will be assessed using the 8-item Morisky Medication Adherence Scale.

SECONDARY OUTCOMES:
Change in HbA1c | Baseline (at recruitment) and 6 months (+/- 4 weeks)
  Part of routine monitoring during doctor's appointment
Change in blood glucose | Baseline (at recruitment) and 6 months (+/- 4 weeks)
  Part of routine monitoring during doctor's appointment
Frequency of dose titrations of oral hypoglycemic agents and insulin | 6 months (+/- 4 weeks) after recruitment
Addition or removal of oral hypoglycemic agents and insulin | 6 months (+/- 4 weeks) after recruitment
Change in health-related quality of life | Baseline (at recruitment) and 6 months (+/- 4 weeks)
  Measured using Audit of Diabetes Dependent Quality of Life - 19 (ADDQoL-19) questionnaire
Change in health status | Baseline (at recruitment) and 6 months (+/- 4 weeks)
  Measured using EuroQol-5D-5L and EuroQol Visual Analogue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Heng McVin Cheen, B.Sc (Pharm), Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore